CLINICAL TRIAL: NCT05113459
Title: A Phase Ⅱ Clinical Study of Disitamab Vedotin Combined With Anti-PD-1 Antibody and Capecitabine in Neoadjuvant Treatment of Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma With Moderate and High Expression of HER2
Brief Title: Disitamab Vedotin Combined With PD-1 and Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancer（RC48-C018）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guoxin Li (Other)
Responsible Party: Sponsor-Investigator, Guoxin Li, Chief Physician, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C018
Record Dates: First submitted 2021-11-02; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Gastric Cancer
Keywords: distamab vedotin PD-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- disitamab vedotin + PD-1+Capecitabine (Experimental): disitamab vedotin：2.5mg/kg,iv,d1,q2w ,6cycle PD-1: 200mg,iv,d1,q2w，6cycle Capecitabine：1000mg/m2 ,po, bid,d1-14,q3w, 4cycle
  Interventions: Drug: Disitamab Vedotin Combined With PD-1 and Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: Disitamab Vedotin Combined With PD-1 and Neoadjuvant Chemotherapy — disitamab vedotin：2.5mg/kg, iv,d1,q2w,6cycle PD-1(Sintilimab ):200mg,iv,d1,q2w,6cycle Capecitabine:1000mg/m2,po,bid,d1-14,q3w,4cycle

SUMMARY:
This trial is a multi-center, open, single-arm, superior phase II clinical study.

DETAILED DESCRIPTION:
The study included 40 patients with gastric cancer or gastroesophageal junction adenocarcinoma with clinical stage T3-4aN+M0; and confirmed after HER2 IHC results Patients with medium and high expression of HER2 (defined as: IHC 2+ 3+); the neoadjuvant treatment plan is: disitamab vedotin + PD-1 + capecitabine; the main goal of the study is to explore The effectiveness of disitamab vedotin combined with PD-1 monoclonal antibody and capecitabine in the neoadjuvant treatment of locally advanced gastric or gastroesophageal junction adenocarcinoma, and ultimately provide a basis for the update of treatment decisions for locally advanced gastric or gastroesophageal junction adenocarcinoma Proof of medical evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form;
2. Age 18-75 years old (including 18 years old and 75 years old);
3. Expected survival period ≥ 12 weeks;
4. ECOG physical fitness score 0 or 1 point;
5. Patients with gastric cancer or gastroesophageal junction adenocarcinoma (Siewert type I-III) confirmed by histology and/or cytology, clinical stage T3-4aN+M0 (determined by the 8th edition of the AJCC staging system);
6. Use pre-treatment endoscopic biopsy samples for HER2 detection in the local laboratory: HER2 high expression confirmed after IHC results (defined as: IHC 2+ 3+);
7. Sufficient organ function:

Bone marrow function: hemoglobin ≥9g/dL; absolute neutrophil count ≥1.5×10 9/L; white blood cell count ≥3.0×10 9/L; platelet ≥100×10 9/L; Liver function: serum total bilirubin ≤1.5 times the upper limit of normal (ULN); when there is no liver metastasis, alanine aminotransferase (ALT), aspartate aminotransferase (AST and alkaline phosphatase (ALP) ≤2.5 × ULN; Renal function: blood creatinine ≤ 1.5×ULN, or creatinine clearance rate (CrCl) ≥ 60 mL/min calculated by Cockcroft-Gault formula method; Heart function: NYHA classification <3; left ventricular ejection fraction ≥50%; 8. For female subjects: women of childbearing age agree to use a medically approved contraceptive method (such as intrauterine device, contraceptives, or contraceptives) during the study treatment period and within 6 months after the end of the study treatment period for the test group participants Set), the blood pregnancy test must be negative within 7 days before the study administration (surgical sterilization or subjects aged ≥60 years can choose not to have a blood pregnancy test), and must be non-lactating; for male subjects: should For surgical sterilization, or agree to use a medically approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period of the experimental group subjects; 9. Must voluntarily join this study and sign an informed consent form.

Exclusion Criteria:

1. Stage IV (metastatic) or unresectable gastric cancer or gastroesophageal junction adenocarcinoma (GEJ) as determined by the investigator;
2. Past systemic treatment for gastric cancer;
3. There is a history of malignant tumors in the 5 years before screening (except for gastric cancer), except for malignant tumors with negligible risk of metastasis or death (for example, 5-year OS rate> 90%), such as cervical carcinoma in situ after appropriate treatment , Non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ or stage I uterine cancer;
4. Severe cardiovascular and cerebrovascular events occurred within 12 months, including but not limited to unstable angina, myocardial infarction, cerebral hemorrhage and cerebral infarction (except for lacunar infarcts that are asymptomatic and do not require treatment);
5. There are other lung diseases that require treatment or are serious, including but not limited to active tuberculosis, interstitial lung disease, etc.;
6. Are suffering from an active infection that requires systemic treatment;
7. There are active autoimmune diseases that require systemic treatment in the past 2 years (such as corticosteroids or immunosuppressive drugs, etc.), and related alternative treatments (such as thyroxine, insulin, or the physiological effects of adrenal or pituitary insufficiency) are allowed Corticosteroid replacement therapy);
8. Major surgery other than diagnosis was received within 4 weeks before the start of study treatment, or major surgery is expected to be required during the study period
9. Serious infections that occurred within 4 weeks before the start of the study treatment, including but not limited to hospitalization due to complications of infection, bacteremia, or severe pneumonia
10. Treat with therapeutic antibiotics within 2 weeks (intravenous antibiotics) or 5 days (oral antibiotics) before starting the study treatment

    - Patients who receive prophylactic antibiotics (for example, to prevent urinary tract infections or prevent exacerbations of chronic obstructive pulmonary disease) are eligible to participate in the study.
11. Have previously received allogeneic stem cell or solid organ transplantation;
12. Any other diseases, metabolic dysfunction, physical examination results or clinical laboratory results that lead to the prohibition of the use of experimental drugs, affect the interpretation of the results, put the patient at a high risk of treatment complications;
13. All treatments using live attenuated vaccines within 4 weeks before the start of the study treatment, or expected to be vaccinated during PD-1 treatment or within 5 months after the last PD-1 administration;
14. Have a clear history or current history of neurological or mental disorders, including epilepsy or dementia;
15. HIV test results are positive; patients with active hepatitis B or C (HBsAg positive and HBV DNA titers higher than the upper limit of normal when HBsAg is positive; HCVAb positive and HCV RNA titers higher than the upper limit of normal when HBsAg is positive);
16. There are factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction;
17. In patients who choose to receive capecitabine, it is required to use the antiviral drug solivudine (antiviral drug) or chemical structure analogs, such as brivudine. These drugs are not allowed to be used within 4 weeks before the start of study treatment including capecitabine;
18. Known to have hypersensitivity or delayed allergic reactions to certain components of RC48-ADC or similar drugs;
19. Those who are allergic to PD-1;
20. It is estimated that the compliance of the patient to participate in this clinical study is sufficient or the researcher thinks that there are other subjects who are not suitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-18 (Estimated); Primary Completion 2023-12-18 (Estimated); Study Completion 2024-06-18 (Estimated)

PRIMARY OUTCOMES:
pathologic Complete Response, PCR | 3 months-6 months
  After completion of neoadjuvant systemic therapy (NAST), hematoxylin and eosin (H&E) assessments were performed on the completely resected gastric cancer or gastroesophageal junction adenocarcinoma sample and all sampled regional lymph nodes. No evidence of residual active tumor cells was found (currently YpT0N0 in the 8th edition of the AJCC staging system)

SECONDARY OUTCOMES:
Major pathologic response, MPR | 3 months-6 months
  Less than 10% of tumor cells were found in pathological resection specimens.
R0 resection rate | 3 months -6 months
  No residue under the microscope after tumor resection
Objective response rate, ORR | 3 months-6 months
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time after neoadjuvant treatment (mainly for solid tumors). It includes complete remission (CR, Complete Response) and partial remission (PR, Partial Response) cases
Relapse-free survival time , RFS | 1-5 years
  The time from the start of randomization to the recurrence of the disease or the death of the patient due to disease progression.
Overall survival , OS | 1-5 years
  The time from the start of randomization to death due to any cause. When the patients who were lost to follow-up before death are recorded, the time of contact with the patient is the last recorded time.

CONTACTS AND LOCATIONS:
Overall Officials: guoxin li, PhD, Principal Investigator — Southern Hospital of Southern Medical University

IPD SHARING:
Plan to Share IPD: No